CLINICAL TRIAL: NCT03629665
Title: Combining Language Therapy With rTMS in Chronic Stage of Aphasia: A Randomized Controlled Trial
Brief Title: Combining Language Therapy With rTMS in Aphasia
Acronym: ILAT+rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paula Heikkinen (Other)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); Aalto University (Other); Freie Universität Berlin (Other)
Responsible Party: Sponsor-Investigator, Paula Heikkinen, Doctoral student, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HelsinkiUniversity/Logopedics
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Aphasia
Keywords: chronic aphasia; rehabilitation; randomized controlled trial (RCT)
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS and naming combined with ILAT (Active Comparator): Interventions: Repetitive navigated Transcranial Magnetic Stimulation, picture naming and Intensive Language Action Therapy
  Interventions: Behavioral: Intensive Language-Action Therapy (ILAT); Device: Repetitive navigated Transcranial Magnetic Stimulation during naming training
- sham rTMS and naming combined with ILAT (Sham Comparator): Interventions: sham Repetitive navigated Transcranial Magnetic Stimulation, picture naming and Intensive Language Action Therapy
  Interventions: Behavioral: Intensive Language-Action Therapy (ILAT)

INTERVENTIONS:
Behavioral: Intensive Language-Action Therapy (ILAT) — ILAT includes communicative language games played in an interactive small-group setting. Three persons with aphasia and one therapist sit around a table and have picture cards in front of them. The card sets include two items of each object or action picture. All participants take turns in making verbal requests. There will be 5 daily sessions (3 hours per session) for two weeks.
Device: Repetitive navigated Transcranial Magnetic Stimulation during naming training — Magnetic stimulation will delivered with a figure-of-eight cooled coil of Navigated Brain Stimulation System during picture naming training. The primary targeted area is the right pars triangularis. In each session, rTMS will be applied at 1-Hz for 20 minutes, 5 daily sessions per week for four weeks.
  Arms: rTMS and naming combined with ILAT

SUMMARY:
With the present RCT, the investigators aimed at finding an optimal protocol for the neurorehabilitation of chronic post-stroke aphasia by combining two promising methods, ILAT (Intensive language action therapy) and 1-Hz rTMS to the right-hemispheric homologue of the anterior language area of Broca (pars triangularis), thus taking advantage of recent research in speech and language sciences, neurorehabilitation and brain research.

DETAILED DESCRIPTION:
New neuromodulation technologies, such as transcranial magnetic stimulation (TMS), are promising tools for neurorehabilitation, aphasia therapy included. Combined with behavioral techniques, Intensive Language-Action Therapy (ILAT), TMS could substantially amplify the beneficial effect of such behavioral therapy alone.

In this randomized study of 17 subjects with post-stroke aphasia in the chronic stage will be studied the combined effect of ILAT and 1-Hz placebo-controlled navigated repetitive TMS (rTMS) to the right-hemispheric inferior frontal cortex (pars triangularis). Participant will be randomized to groups A and B. Participants in group A will receive a 2-week period of rTMS during naming training where they name pictures every ten second displayed on the screen, followed by 2-weeks of rTMS and naming combined with ILAT. Those in group B will receive the same behavioral therapy but TMS is replaced by sham stimulation.

Language performance will be measured before, during and after the interventions for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* presence of a single clinically documented stroke
* chronic stage (at least 12 months post-stroke)
* aphasia documented using the WAB test
* no recurring utterances or severe global (total) aphasia
* residual ability to understand simple task instructions
* availability of information about medication
* right-handedness
* native speakers of Finnish.

Exclusion Criteria:

* severe global (total) aphasia (Boston naming test less 3 points)
* neglect, agnosia, severe vision impairment or hearing loss
* severe attention or memory deficits
* left-handedness
* cardiac pacemaker or other stimulators
* diagnosis of severe diabetes or severe depression
* additional neurological diagnoses
* other interventions, including speech therapy, in the same time period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-01 (Actual)

PRIMARY OUTCOMES:
The Western Aphasia Battery | Change in AQ performed at weeks 1 (baseline), 4 and 7 and follow up 3 months after therapy completion
  aphasia quotient (AQ) measurement

SECONDARY OUTCOMES:
The Boston naming test | Change in picture naming ability between weeks 1 (baseline), 4 and 7 and follow up 3 months after therapy completion
  picture naming ability
The Action naming test | Change in picture naming ability between weeks 1 (baseline), 4 and 7 and follow up 3 months after therapy completion
  picture naming ability

CONTACTS AND LOCATIONS:
Overall Officials: Anu Klippi, Professor, Principal Investigator — University of Helsinki; Jyrki Mäkelä, MD, Study Chair — BioMag Laboratory, Helsinki University Hospital; Friedemann Pulvermüller, Professor, Study Chair — Brain Language Laboratory, Department of Philosophy and Humanities, WE4, Freie Universität Berlin; Risto Ilmoniemi, Professor, Study Chair — Department of Neuroscience and Biomedical Engineering, Aalto University School of Science

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heikkinen PH, Pulvermuller F, Makela JP, Ilmoniemi RJ, Lioumis P, Kujala T, Manninen RL, Ahvenainen A, Klippi A. Combining rTMS With Intensive Language-Action Therapy in Chronic Aphasia: A Randomized Controlled Trial. Front Neurosci. 2019 Feb 4;12:1036. doi: 10.3389/fnins.2018.01036. eCollection 2018. PMID 30778280